CLINICAL TRIAL: NCT00557830
Title: Randomized Phase IIb Study of Sorafenib Dose Escalation in Patients With Previously Untreated Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Randomized Study of Sorafenib Dose Escalation in Patients With Previously Untreated Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to enrollment when it became clear that enrollment was too slow to complete the full enrollment target within the time frame allowed.
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVJARCC0702
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Escalated Dose (Active Comparator): Eligible patients will be randomized 2:1 to either Group A (escalated dose regimen) or Group B (standard dose regimen). Patients randomized to Group A will receive sorafenib 600 mg bid for Weeks 5 through 8 (Dose Level 2). Patients who tolerate this dose through Week 8 will be further escalated to Dose Level 3 (800 mg po bid) for Weeks 9 through 12.
  Interventions: Drug: Sorafenib Escalated Dose
- Group B: Standard Dose (Active Comparator): Eligible patients will be randomized 2:1 to either Group A (escalated dose regimen) or Group B (standard dose regimen). Patients randomized to Group B will receive Dose Level 1 (sorafenib 400 mg po bid) until progression of disease, intolerable toxicity, patient refusal to continue with the study, or investigator decision to remove the patient from the study.
  Interventions: Drug: Sorafenib Standard Dose

INTERVENTIONS:
Drug: Sorafenib Escalated Dose — Patients randomized to Group A will receive sorafenib 600 mg bid for Weeks 5 through 8 (Dose Level 2). Patients who tolerate this dose through Week 8 will be further escalated to Dose Level 3 (800 mg po bid) for Weeks 9 through 12.
  Other Names: Nexavar
  Arms: Group A: Escalated Dose
Drug: Sorafenib Standard Dose — Patients randomized to Group B will receive Dose Level 1 (sorafenib 400 mg po bid) until progression of disease, intolerable toxicity, patient refusal to continue with the study, or investigator decision to remove the patient from the study.
  Other Names: Nexavar
  Arms: Group B: Standard Dose

SUMMARY:
The primary objective of this study is to compare the effectiveness of a dose-escalation regimen (400 to 800mg bid) relative to the standard dosing regimen (400mg bid) of sorafenib given in patients with metastatic RCC.

The secondary objectives are to evaluate the effects of the dose-escalation regimen on the quality of life (QoL) of patients with metastatic RCC and to characterize the safety and tolerability profile of a dose-escalation regimen of sorafenib in patients with metastatic RCC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Diagnosis of unresectable/metastatic renal cell carcinoma (RCC). Nonclear cell histology is permitted (except for medullary, collecting duct, or sarcomatoid >50% of specimen). Prior metastasectomy is permitted as long as there is measurable disease at time of consent.
* Karnofsky Performance Status of 50% or greater at study entry.
* Adequate bone marrow, liver and renal function as assessed by the following: o Hemoglobin ≥ 9.0 g/dL. o ANC ≥ 1500/mm3. o Platelet count ≥ 100,000/mm3. o Total bilirubin ≤ 1.5 ULN. o ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver involvement). o Creatinine ≤ 1.5 × ULN.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and sexually active men must agree to use adequate barrier contraception prior to study entry, for the duration of study participation, and for at least three months after the last administration of sorafenib.
* INR < 1.5 or a PT/ PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Prior systemic anticancer treatment for metastatic disease, including investigational therapy.
* Prior treatment with bevacizumab, sunitinib, or sorafenib even in the adjuvant setting.
* Prior cytokine therapy with interleukin (IL)-2 or interferon (IFN) for metastatic disease.
* Active malignancy other than RCC (except non-melanoma skin cancer) within 5 years of enrollment.
* Hemodialysis or peritoneal dialysis.
* Treatment with radiotherapy within 2 weeks of enrollment.
* Cardiac disease: Congestive heart failure Class II or higher per NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Uncontrolled CNS metastases. All patients must undergo a CT) scan/MRI of the brain to exclude brain metastasis. Patients with adequately treated CNS disease may be considered for participation as long as the first dose of sorafenib is 4 weeks after completion of CNS therapy.
* Uncontrolled hypertension defined as SBP > 150 mmHg or DBP > 90 mmHg, despite optimal medical management.
* Active clinically serious infection > Grade 2 per the CTCAE v3.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ Grade 2 per CTCAE v3.0 within 4 weeks of administration of the first dose of study drug.
* Any other hemorrhage/bleeding event ≥ Grade 3 per CTCAE v3.0 within 4 weeks of administration of the first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of administration of the first study drug dose.
* Use of St. John's Wort, rifampin (rifampicin), phenytoin, Phenobarbital, carbamazepine, dexamethasone.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Assikis, MD, Principal Investigator — Acorn Cardiovascular, Inc.
Locations (13):
- United States (13):
  - Clopton Clinic, Jonesboro, Arkansas
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Advanced Medical Specialties, Miami, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Peachtree Hematology Oncology Consultants, Atlanta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Mid-Illinois Hematology and Oncology Associates, Ltd., Normal, Illinois
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Gaston Hematology and Oncology, Gastonia, North Carolina
  - Pacific Oncology, PC, Beaverton, Oregon
  - The Lancaster Cancer Center, Ltd, Lancaster, Pennsylvania
  - The West Clinic, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 community oncology sites across the US associated with the ACORN network participated in this study. Enrollment started in January 2008 and was closed in August 2008 due to the low rate of accrual and lack of funds beyond the current level of support from Bayer.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening phase that could last up to 4 weeks during which pre-study assessments were completed. Eligible subjects then underwent a screening treatment phase in which they received commercial sorafenib for 4 weeks.
Groups:
- Screening Treatment Phase: After patients have signed informed consent and found to be eligible they will be started on standard dose sorafenib (800 mg/d) which constitutes the screening treatment phase. Patients who have been receiving treatment with commercial sorafenib outside of a clinical trial for < 2 weeks may also be able to participate in this trial provided all screening/baseline procedures are completed. During the screening treatment phase, commercial sorafenib will be prescribed. A patient will be eligible for randomization if (s)he successfully receives treatment with sorafenib for 4 weeks at 400 mg (po) bid (Study Weeks 1 through 4).
- Group A: Escalated Dose: Eligible patients will be randomized 2:1 to either Group A (escalated dose regimen) or Group B (standard dose regimen). Patients randomized to Group A will receive sorafenib 600 mg bid for Weeks 5 through 8 (Dose Level 2). Patients who tolerate this dose through Week 8 will be further escalated to Dose Level 3 (800 mg po bid) for Weeks 9 through 12.
  Sorafenib Escalated Dose :
  Patients randomized to Group A will receive sorafenib 600 mg bid for Weeks 5 through 8 (Dose Level 2). Patients who tolerate this dose through Week 8 will be further escalated to Dose Level 3 (800 mg po bid) for Weeks 9 through 12.
- Group B: Standard Dose: Eligible patients will be randomized 2:1 to either Group A (escalated dose regimen) or Group B (standard dose regimen). Patients randomized to Group B will receive Dose Level 1 (sorafenib 400 mg po bid) until progression of disease, intolerable toxicity, patient refusal to continue with the study, or investigator decision to remove the patient from the study.
  Sorafenib Standard Dose :
  Patients randomized to Group B will receive Dose Level 1 (sorafenib 400 mg po bid) until progression of disease, intolerable toxicity, patient refusal to continue with the study, or investigator decision to remove the patient from the study.
Period: Screening Treatment Phase
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Started | 12 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Unable to tolerate standard dose | 3 | 0 | 0
Period: Treatment Phase
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Started | 0 | 4 | 2
Completed | 0 | 4 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose | Total
Number analyzed (Participants) | 12 | 4 | 2 | 18
Age Continuous [Mean (Standard Deviation); unit: years]
  Screening Treatment Phase | 62.2 (10.99) | NA (NA) — Age for screening population only | NA (NA) — Age for screening population only. | 62.2 (10.99)
  Randomization Phase | NA (NA) — Age for randomization population only. | 66.0 (6.38) | 58.5 (7.78) | 63.5 (7.18)
Sex/Gender, Customized [Number; unit: Participants]
  Female (Screening Treatment Phase) | 3 | 0 | 0 | 3
  Male (Screening Treatment Phase) | 9 | 0 | 0 | 9
  Female (Randomization Phase) | 0 | 2 | 0 | 2
  Male (Randomization Phase) | 0 | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | NA — See Customized Region of Enrollment Table | NA — See Customized Region of Enrollment Table | NA — See Customized Region of Enrollment Table | 0
Region of Enrollment, Customized [Number; unit: participants]
  United States (Screening Treatment Phase) | 12 | NA — Region for randomization population only | NA — Region for randomization population only | 12
  United States (Randomization Phase) | NA — Region for screening population only | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR + PR) Determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria.
Description: Response was evaluated via changes from baseline in radiological tumor measurements performed every 8 weeks and at the end of treatment unless clinically indicated prior to that. Confirmatory scans were to be obtained no less than 4 weeks but no more than 6 weeks following initial documentation of objective response. Response was evaluated using RECIST criteria, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease; Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions or the appearance of one or more new lesions.
Time Frame: Overall response will be measured at baseline and every 8 weeks , unless clinically indicated prior to that, until the end of treatment.
Measure: Number; unit: Participants
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Number analyzed (Participants) | 0 | 4 | 2
Participants
  Complete Response (CR) |  | 0 | 0
  Partial Response (PR) |  | 0 | 0
  Stable Disease (SD) |  | 3 | 1
  Progressive Disease (PD) |  | 1 | 1

2. Secondary Outcome: PFS Rate at 9, 13 and 17 Months
Description: Due to the early study closure and the small sample size, the PFS rate at 9, 13, and 17 months were not evaluated.
Time Frame: PFS was to be measured at 9, 13, and 17 months.
Population: Due to the early study closure and the small sample size, the PFS rate at 9, 13, and 17 months were not evaluated.
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Survival Rate
Description: Due to the early study closure and the small sample size, overall survival rate was not evaluated.
Time Frame: Overall survival was measured from day 1 of treatment until the end of treatment and then every 4 months thereafter until death.
Population: Due to the early study closure and the small sample size, overall survival rate was not evaluated.
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Changes From Baseline in Symptom Burden
Description: The Patient Care Monitor Version 2.0 (PCM) is an tablet computer based assessment system that measures patient reported outcomes (PROs) in medical patients with a particular emphasis on symptoms related to cancer and its treatment.
  The PCM comprises 86 items which include 8 items answered only by females (e.g. menstrual cramping). Each item is presented so that the patient rates the degree to which the item has been a problem in the past week (0 not a problem to 10 as bad as possible).
Time Frame: The PCM was administered during screening, at each scheduled visit (approximately every 4 weeks), and at the end of treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Number analyzed (Participants) | 12 | 4 | 2
units on a scale
  Hives (Welts)-Baseline | 0 (0) | 0 (0) | 0 (0)
  Hives (Welts)-Post-BL | 1.2 (2.94) | 0.2 (0.38) | 0 (0)
  Sinus Problem-Baseline | 1.1 (2.51) | 2.3 (3.86) | 0 (0)
  Sinus Problem-Post-BL | 1.1 (1.89) | 2.4 (2.54) | 0.1 (0.11)
  Chest Pain-Baseline | 0.1 (0.32) | 0.3 (0.5) | 0 (0)
  Chest Pain-Post-BL | 0.3 (0.56) | 0.4 (0.54) | 0 (0)
  Rapid Heart Beat-Baseline | 0.8 (2.53) | 2 (4) | 0 (0)
  Rapid Heart Beat-Post-BL | 0.3 (0.75) | 0.9 (1.2) | 0 (0)
  Swelling-Baseline | 0.3 (0.95) | 0.8 (1.5) | 0 (0)
  Swelling-Post-BL | 1 (2.28) | 0 (0.06) | 0 (0)
  Constitutional Chills-Baseline | 0.2 (0.63) | 0.5 (1) | 0 (0)
  Constitutional Chills-Post-BL | 0.9 (1.69) | 0.8 (1.32) | 0 (0)
  Fatigue-Baseline | 2.3 (2.54) | 3.8 (3.3) | 2 (2.83)
  Fatigue-Post-BL | 2.7 (2.72) | 5 (3.22) | 0.5 (0.71)
  Fever-Baseline | 0.4 (1.26) | 1 (2) | 0 (0)
  Fever-Post-BL | 0.9 (1.47) | 1.4 (2) | 0 (0)
  Weight Gain-Baseline | 1.3 (2.75) | 1.8 (3.5) | 0 (0)
  Weight Gain-Post-BL | 0.3 (0.78) | 0 (0) | 0 (0)
  Weight Loss-Baseline | 0.4 (1.26) | 1 (2) | 0 (0)
  Weight Loss-Post-BL | 0.7 (1.39) | 1.6 (2.14) | 0 (0)
  Change In Taste-Baseline | 0.5 (1.27) | 1 (2) | 0 (0)
  Change In Taste-Post-BL | 0.8 (1.41) | 2.2 (1.81) | 0 (0)
  Difficulty Hearing-Baseline | 0.7 (2.21) | 1.8 (3.5) | 0 (0)
  Difficulty Hearing-Post-BL | 0.5 (1.24) | 0 (0) | 0 (0)
  Dry Mouth-Baseline | 0.8 (2.04) | 0 (0) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Dry Mouth-Post-BL | 1.7 (1.5) | 2 (1.7) | 2.7 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Mouth Sores/Ulcers-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Mouth Sores/Ulcers-Post-BL | 0.9 (1.53) | 0.6 (1.04) | 0 (0)
  Sore Throat-Baseline | 0 (0) | 0 (0) | 0 (0)
  Sore Throat-Post-BL | 0.4 (0.63) | 0.5 (0.54) | 0 (0)
  Trouble Swallowing-Baseline | 0 (0) | 0 (0) | 0 (0)
  Trouble Swallowing-Post-BL | 0.3 (0.62) | 0.3 (0.5) | 0 (0)
  Day Sweat-Baseline | 0 (0) | 0 (0) | 0 (0)
  Day Sweat-Post-BL | 0 (0) | 0 (0) | 0 (0)
  Hot Flashes/Flushes-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Hot Flashes/Flushes-Post-BL | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Night Sweat-Baseline | 1.7 (3.65) | 4.3 (5.06) | 0 (0)
  Night Sweat-Post-BL | 0.4 (1.3) | 1.1 (2.25) | 0 (0)
  Reduced Sexual Enjoyment-Baseline | 0.2 (0.63) | 0 (0) | 0 (0)
  Reduced Sexual Enjoyment-Post-BL | 0.4 (1.08) | 0.9 (1.75) | 0 (0)
  Dry Eyes-Baseline | 0.7 (2) | 1.5 (3) | 0 (0)
  Dry Eyes-Post-BL | 0.9 (1.49) | 1.4 (1.79) | 0 (0)
  Tearing-Baseline | 1.1 (1.96) | 2.3 (2.63) | 0 (0)
  Tearing-Post-BL | 0.5 (1.36) | 1.2 (2.35) | 0 (0)
  Trouble Seeing-Baseline | 0.4 (1.33) | 1 (2) | 0 (0)
  Trouble Seeing-Post-BL | 1.6 (2.9) | 2 (3.37) | 0 (0)
  Constipation-Baseline | 0.1 (0.32) | 0.3 (0.5) | 0 (0)
  Constipation-Post-BL | 0.2 (0.45) | 0.5 (0.71) | 0.3 (0.35)
  Decrease in Appetite-Baseline | 0 (0) | 0 (0) | 0 (0)
  Decrease in Appetite-Post-BL | 0.8 (1.89) | 2.4 (2.87) | 0 (0)
  Diarrhea-Baseline | 0 (0) | 0 (0) | 0 (0)
  Diarrhea-Post-BL | 0.8 (0.88) | 1.1 (0.77) | 1.3 (1.88)
  Heartburn-Baseline | 0.7 (1.25) | 1.3 (1.89) | 0 (0)
  Heartburn-Post-BL | 1.2 (1.67) | 2.7 (2.17) | 0 (0)
  Increase in Appetite-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Increase in Appetite-Post-BL | 0.2 (0.48) | 0.1 (0.14) | 0 (0)
  Nausea-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Nausea-Post-BL | 0.8 (1.11) | 1.4 (1.53) | 0.5 (0.71)
  Vomiting-Baseline | 0 (0) | 0 (0) | 0 (0)
  Vomiting-Post-BL | 0.4 (0.86) | 1.1 (1.31) | 0 (0)
  Menstrual Pain/Cramping-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Menstrual Pain/Cramping-Post-BL | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Problem with Urination-Baseline | 0.5 (1.08) | 1.3 (1.5) | 0 (0)
  Problem with Urination-Post-BL | 0.2 (0.48) | 0 (0) | 0 (0)
  Vaginal Bleeding-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Vaginal Bleeding-Post-BL | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Vaginal Discharge-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Vaginal Discharge-Post-BL | 0.1 (0.14) | 0.1 (0.18) | NA (NA) — All subjects in Group B are male.
  Vaginal Dryness-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Vaginal Dryness-Post-BL | 0 (0.07) | 0.1 (0.09) | NA (NA) — All subjects in Group B are male.
  Vaginal Itching-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Vaginal Itching-Post-BL | 0.5 (0.51) | 0.2 (0.27) | NA (NA) — All subjects in Group B are male.
  Bleeding-Baseline | 0.2 (0.63) | 0 (0) | 0 (0)
  Bleeding-Post-BL | 0.1 (0.17) | 0.1 (0.25) | 0 (0)
  Bruising-Baseline | 0.2 (0.63) | 0 (0) | 0 (0)
  Bruising-Post-BL | 0.4 (1.35) | 0 (0) | 0 (0)
  New Lump/Mass-Baseline | 0 (0) | 0 (0) | 0 (0)
  New Lump/Mass-Post-BL | 0.2 (0.79) | 0.7 (1.38) | 0 (0)
  Breast Tenderness-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Breast Tenderness-Post-BL | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Dry Skin-Baseline | 1.4 (2.99) | 2 (4) | 3 (4.24)
  Dry Skin-Post-BL | 2.5 (3.34) | 3.2 (2.72) | 0.2 (0.33)
  Hair Loss-Baseline | 0 (0) | 0 (0) | 0 (0)
  Hair Loss-Post-BL | 1.2 (1.86) | 3.3 (1.9) | 0.5 (0.65)
  Itching-Baseline | 1.1 (2.33) | 1.3 (2.5) | 3 (4.24)
  Itching-Post-BL | 1.7 (2.78) | 1.2 (0.85) | 0.1 (0.19)
  Nails Change-Baseline | 0 (0) | 0 (0) | 0 (0)
  Nails Change-Post-BL | 0.7 (1.27) | 1.9 (1.62) | 0.1 (1.6)
  Nipple Discharge-Baseline | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Nipple Discharge-Post-BL | 0 (0) | 0 (0) | NA (NA) — All subjects in Group B are male.
  Rash-Baseline | 0 (0) | 0 (0) | 0 (0)
  Rash-Post-BL | 1.7 (3) | 1.1 (2.09) | 0 (0)
  Joint Pain-Baseline | 1 (2.16) | 1 (2) | 0 (0)
  Joint Pain-Post-BL | 1.3 (2.14) | 0.9 (1.06) | 0 (0)
  Muscle Aches-Baseline | 0.5 (1.08) | 0.5 (1) | 0 (0)
  Muscle Aches-Post-BL | 1.2 (2.06) | 0.8 (0.99) | 0.3 (0.35)
  Weakness of Body Parts-Baseline | 0.6 (1.07) | 1 (1.41) | 0 (0)
  Weakness of Body Parts-Post-BL | 1.8 (2.3) | 4 (2.74) | 0 (0)
  Burning Sensation in Hands or Feet-Baseline | 0.8 (1.93) | 2 (2.83) | 0 (0)
  Burning Sensation in Hands or Feet-Post-BL | 2.3 (3.12) | 2.6 (2.62) | 0 (0)
  Daytime Sleepiness-Baseline | 0.5 (0.97) | 0.8 (1.5) | 0 (0)
  Daytime Sleepiness-Post-BL | 1.1 (1.52) | 1.9 (1.91) | 0 (0)
  Dizziness/Lightheadedness-Baseline | 0.2 (0.42) | 0.5 (0.58) | 0 (0)
  Dizziness/Lightheadedness-Post-BL | 0.4 (0.68) | 0.8 (0.78) | 0 (0)
  Memory Loss-Baseline | 0 (0) | 0 (0) | 0 (0)
  Memory Loss-Post-BL | 0.3 (0.87) | 0 (0) | 0 (0)
  Numbness/Tingling-Baseline | 0 (0) | 0 (0) | 0 (0)
  Numbness/Tingling-Post-BL | 0.7 (1.35) | 0.2 (0.19) | 0 (0)
  Trouble Sleeping at Night-Baseline | 1.3 (2.06) | 1 (2) | 3 (4.24)
  Trouble Sleeping at Night-Post-BL | 1.6 (1.81) | 2.5 (2.28) | 1 (1.41)
  Trouble Thinking-Baseline | 0 (0) | 0 (0) | 0 (0)
  Trouble Thinking-Post-BL | 0 (0.14) | 0.1 (0.25) | 0 (0)
  Headache-Baseline | 0.1 (0.32) | 0.3 (0.5) | 0 (0)
  Headache-Post-BL | 0.5 (0.6) | 0.7 (0.55) | 0 (0)
  Pain-Baseline | 0.8 (1.14) | 1.3 (1.5) | 0 (0)
  Pain-Post-BL | 2 (2.51) | 2.6 (2.13) | 0 (0)
  Attend Paid Job-Baseline | 1.1 (2.42) | 2 (3.37) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Attend Paid Job-Post-BL | 3.8 (3.98) | 3.7 (3.56) | 0 (0)
  Attend Social Activity-Baseline | 0.6 (1.67) | 1.3 (2.5) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Attend Social Activity-Post-BL | 1.8 (2.56) | 3 (2.68) | 0 (0)
  Bathe or Dress-Baseline | 0.2 (0.67) | 0.5 (1) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Bathe or Dress-Post-BL | 1.3 (1.81) | 1.4 (1.69) | 0 (0)
  Cook for Self-Baseline | 0.8 (2.33) | 1.8 (3.5) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Cook for Self-Post-BL | 1.6 (2.45) | 2.6 (2.67) | 0 (0)
  Driving-Baseline | 0.3 (1) | 0.8 (1.5) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Driving-Post-BL | 1.2 (1.68) | 2.2 (2.09) | 0 (0)
  Function Normally-Baseline | 2.3 (3.2) | 3.8 (4.35) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Function Normally-Post-BL | 2.9 (2.8) | 3.8 (2.88) | 0 (0)
  Hard Work or Activity-Baseline | 2.3 (2.87) | 1.3 (1.15) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Hard Work or Activity-Post-BL | 3.9 (3.1) | 5.3 (3.52) | 0 (0)
  Household Work-Baseline | 1.6 (2.35) | 2.3 (3.3) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Household Work-Post-BL | 2.8 (2.29) | 4.2 (2.84) | 0 (0)
  Light Work or Activity-Baseline | 0.6 (1.13) | 0 (0) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Light Work or Activity-Post-BL | 2.6 (2.36) | 3.4 (2.65) | 0 (0)
  Run-Baseline | 2 (2.98) | 0.7 (1.15) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Run-Post-BL | 3.8 (3.96) | 5.9 (3.97) | 0 (0)
  Run Errands-Baseline | 1.7 (3.32) | 3.8 (4.35) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Run Errands-Post-BL | 2.5 (3) | 4.6 (3.73) | 0 (0)
  Sit Up-Baseline | 0.2 (0.67) | 0.5 (1) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Site Up-Post-BL | 0 (0.14) | 0.1 (0.25) | 0 (0)
  Stay Out of Bed-Baseline | 0.2 (0.67) | 0.5 (1) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Stay Out of Bed-Post-BL | 0.5 (1.11) | 1.1 (1.66) | 0 (0)
  Walk-Baseline | 0.8 (1.72) | 0.5 (1) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Walk-Post-BL | 3.1 (3.19) | 3.4 (2.26) | 0 (0)
  Crying/Feeling Like Crying-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Crying/Feeling Like Crying-Post-BL | 0.2 (0.46) | 0.2 (0.36) | 0 (0)
  Feeling Guilty-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Feeling Guilty-Post-BL | 0.2 (0.72) | 0 (0) | 0 (0)
  Feeling Helpless-Baseline | 0 (0) | 0 (0) | 0 (0)
  Feeling Helpless-Post-BL | 0.4 (0.94) | 0.8 (1.5) | 0 (0)
  Feeling Hopeless-Baseline | 0 (0) | 0 (0) | 0 (0)
  Feeling Hopeless-Post-BL | 0.1 (0.43) | 0.4 (0.75) | 0 (0)
  Feeling I Would Be Better Off Dead-Baseline | 0 (0) | 0 (0) | 0 (0)
  Feeling I Would Be Better Off Dead-Post-BL | 0.2 (0.47) | 0.2 (0.38) | 0 (0)
  Feeling Worthless-Baseline | 0 (0) | 0 (0) | 0 (0)
  Feeling Worthless-Post-BL | 0.3 (0.69) | 0.6 (1.13) | 0 (0)
  Lost Interest in People-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Lost Interest in People-Post-BL | 0.4 (1.03) | 0.6 (1.13) | 0 (0)
  Lost Interest in Pleasurable Activities-Baseline | 0.1 (0.32) | 0 (0) | 0 (0)
  Lost Interest in Pleasurable Activities-Post-BL | 0.5 (1.3) | 1.4 (2.14) | 0 (0)
  Nervous, Tense, Anxious-Baseline | 1 (1.25) | 0.8 (0.96) | 1.5 (2.12)
  Nervous, Tense, Anxious-Post-BL | 0.6 (0.87) | 0.9 (1.15) | 0 (0)
  Sad (Depressed)-Baseline | 0 (0) | 0 (0) | 0 (0)
  Sad (Depressed)-Post-BL | 0.5 (0.95) | 0.6 (1.25) | 0 (0)
  Worry-Baseline | 1 (1.25) | 0.8 (0.96) | 1.5 (2.12)
  Worry-Post-BL | 0.6 (1.05) | 0.8 (1.06) | 0 (0)
  Coughing-Baseline | 1.6 (2.95) | 2 (4) | 3 (4.24)
  Coughing-Post-BL | 1 (2.29) | 2.4 (3.79) | 0 (0)
  Shortness of Breath-Baseline | 2.2 (2.86) | 3.3 (3.59) | 0 (NA) — Only one subject provided a response at this timepoint; therefore, there is no SD.
  Shortness of Breath-Post-BL | 2.1 (2.7) | 4 (3.47) | 0 (0)
  Wheezing-Baseline | 1.2 (2.57) | 2 (4) | 0.5 (0.71)
  Wheezing-Post-BL | 1 (2.29) | 2 (3.62) | 0 (0)

5. Post Hoc Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. Progression is defined per RECIST criteria as at least a 20% increase in the sum of the longest dimension (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new non-target lesions and/or unequivocal progression of existing non-target lesions. The median progression free survival is the parameter used to describe PFS.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed every 8 weeks) or death, whichever occurred first
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Number analyzed (Participants) | 12 | 4 | 2
Months | 11.37 [2.83 to 17.35] | 5.77 [2.83 to 7.56] | NA [11.17 to NA] — Only 1 survival even occurred for Group B.

ADVERSE EVENTS:
Time Frame: Adverse events were collected when the patient began taking sorafenib until one month after the end of study treatment.
Description: Systematic assessment- subjects were assessed for adverse events every 4 weeks by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Screening Treatment Phase | Group A: Escalated Dose | Group B: Standard Dose
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/4 | 0/2
Other Adverse Events (participants affected / at risk) | 12/12 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Treatment Phase (N=12) | Group A: Escalated Dose (N=4) | Group B: Standard Dose (N=2)
Bronchitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Treatment Phase (N=12) | Group A: Escalated Dose (N=4) | Group B: Standard Dose (N=2)
Eye irritation (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Stomatitis (General disorders) | 3 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Blood amylase increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 2 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The decision to close the study was made by the funder , Bayer HealthCare Pharmaceuticals, in collaboration with ACORN due to the low rate of accrual in light of study timelines and the lack of funds beyond the current level of support from Bayer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation of Sponsored Research results, Researcher agrees to provide Bayer with such presentation, abstract, or manuscript at least 30 days prior to its presentation or submission for the sole purpose of allowing Bayer to redact confidential information and protect any existing or future patients. The Principal Investigator shall acknowledge Bayer contributions where appropriate.